CLINICAL TRIAL: NCT01063530
Title: Effects of DIammine SIlver Fluoride Placed Over Cervical Lesions of Permanent Teeth to Reduce Tooth Sensitivity
Brief Title: Effects of DIammine SIlver Fluoride on Tooth Sensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: University of Washington (Other)
Responsible Party: Jorge L Castillo, Universidad Peruana Cayetano Heredia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0000054110
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Dental Sensitivity; Gingival Condition
Keywords: FLuoride; Dental Sensitivity; Abfraction; Cervical lesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diammine Silver Fluoride (Experimental): Application fo diammine silver fluoride in cervical lesions
  Interventions: Device: DIammine SIlver fluoride
- Distilled water (Placebo Comparator): Application of distilled water in cervical lesions
  Interventions: Device: DIstilled water

INTERVENTIONS:
Device: DIammine SIlver fluoride — Application of Diammine SIlver Fluoride in cervical lesions
  Arms: Diammine Silver Fluoride
Device: DIstilled water — Application of distilled water in cervical lesions
  Arms: Distilled water

SUMMARY:
The purpose of the study is to confirm the clinical effectiveness and safety of topical diammine silver fluoride (DASF) as a tooth desensitizer in adulst by comparing it to the application of sterile water.

The study will be conducted in two different sites in Peru. Participantes will be 144 adults who will have at least one vital maxillary or mandibular cuspid or premolar with a cervical defect on the buccal surface and clinical hypersensitivity in response to air. Subjects will be randomly assigned to a topical application of DAS or sterile water.

The reduction of pain (sensitivity) using a 100 mm VAS, will be determined. Safety will be also determined by evaluating the gingival condition (erythema, white changes, ulceration, staining) before and ater the application of the products. The evaluation times will be 24 hours and 7 days.

DETAILED DESCRIPTION:
Specific Aim: The purpose of this study is to confirm the clinical effectiveness and safety of topical diammine silver fluoride (DASF) as a tooth desensitizer in adults by comparing it to the application of sterile water.

Design: This is a blinded, randomized clinical trial with two groups. The study will be 1 week in duration.

Study Sites: The study will be conducted in two different sites in Peru (Cayetano University and Universidad Andina del Cusco). Cayetano University is a major private university in South America. It is a recipient of Fogerty International Center funds from NIH and has a history of successful collaboration with US universities, including the University of Washington. Dr. Castillo, the principal investigator, received his training in orthodontics at the University of Washington and is familiar with US clinical trials procedures.

Subjects: Participants will be 144 adults (18 to 50 years). Males and females will be included. Each site (Cayetano and Cusco) will recruit 72 subjects.

Inclusion Criteria: To be included the subject must have at least one vital maxillary or mandibular cuspid or premolar with a cervical defect on the buccal surface and clinical hypersensitivity in response to air with a score not less than 15 on the VAS for pain (described below). The individual will have generally healthy gum tissue surrounding this tooth and no ulceration, and no leukoplakia (white changes) in this gingival tissue.

Exclusion Criteria: Excluded will be subjects who are using any type of commercially available tooth desensitizer, have received a fluoride varnish treatment within the last month, or who are taking prescription medications of any kind, are taking aspirin or nonsteroidal anti-inflammatory drugs habitually, and women who are pregnant. Individuals using smokeless tobacco will be excluded. Individuals with known sensitivity to silver or other heavy-metal ions will be excluded.

Subject Recruitment: Subjects will be recruited from the patient populations of Cayetano University School of Dentistry and Universidad Andina del Cusco School of Dentistry. Subjects will be offered a small financial incentive for participation, paid as $10 US at the second visit (24 hours) and $20 US at the 1-week check.

Protection of Human Subjects: The Institutional Review Board of Cayetano University will review the protocol, and the informed consent of all participants will be obtained. The Cayetano IRB is familiar with US procedures because NIH level work is conducted there.

Treatment Conditions: Subjects will be randomly assigned to a topical application of DASF or sterile water. The randomization will be stratified on study site and baseline sensitivity score to a 5-second blast of pressurized air at 2 cm distance from the tooth (see description of measures below). Odor is not a threat to blinding because the smell is not detectable clinically when using such small quantities. Taste is not a threat in this study because only mg amounts of material are applied, and the tooth is air-dried after application.

The random treatment assignments will be generated by the project statistician. The randomization to the two treatments will be done with stratification on study site and baseline pain score (<37 and ≥37), and blocking to ensure the two treatment groups will be balanced across the study period and within each stratum. The stratification at 37 was chosen from the literature (Ritter et al., 2006, paper appended) to ensure balance. A pretest of the VAS with 10 pretest subjects in Peru confirmed that the mean response was in this range. Block sizes will be equal to 2 or 4, and will be chosen randomly with 2/3 and 1/3 probability, respectively. The randomization list will be prepared using the "sample" function of R statistical software (Version 2.7.1, The R Foundation for Statistical Computing, 2008). The assignments will be recorded on slips of paper numbered consecutively within each stratum and then placed inside sealed envelopes sequentially numbered by stratum. The statistician will retain the master list, and the code will not be broken until all the data are analyzed. The clinician will open the envelope and apply the agent. The agents (active or control) will be packaged in identical bottles labeled as A or B. The packaging will be done by the investigational pharmacy at Cayetano University.

Diammine silver fluoride (Saforide, Toyo Seiyaku Kasei Co. Ltd. Osaka, Japan) will be used. Saforide is a clear and colorless liquid with a weak odor of ammonia. It is a solution of diammine silver fluoride [Ag(NH3)2F]. It includes not less than 24.4w/v% and not more than 26.8 w/v% of silver (Ag), not less than 5.0 w/v% and not more than 5.9 w/v% of fluorine (F).

Measures:

Primary Outcome-Clinical Reduction of pain (sensitivity)-The teeth will be isolated with cotton gauze, and subjects will report tooth pain on a 100-mm VAS (Ritter et al., 2006, paper appended) before treatment and after treatment to a 5-second blast of pressurized air at 2 cm distance from the tooth. The VAS will be anchored with "no pain" and "intolerable pain." The follow-up test will be repeated at 24 hours and 1 week later.

The assessment will be conducted in Spanish (forms appended). We have pretested the scale to be sure the descriptors are translated properly. The terms "sensitivity," "dentin sensitivity" and "pain" are used interchangeably in this literature. For subjects with multiple test teeth, VAS scores will be averaged to produce one score per subject at each time point. The primary end-point will be 1 week after treatment.

The study will test application of diammine silver fluoride in a single visit because previous work shows that a single application physically blocks most dentinal tubules and that additional applications are not necessary, as sensitivity is reduced significantly. The clinical procedure is that a disposable microbrush is dipped into a small drop of the diammine silver fluoride or the control and then applied to the surface for 1 second, as is done clinically. Then the surface is gently air-dried and the procedure repeated.

Safety Damage to Gingiva-Tissues will be photographed before application of any agents to establish the normal baseline condition. Gingival tissues surrounding each tooth treated will be examined clinically immediately after treatment, at 24 hours and one week later. A photograph of the assignment envelope and ID will be taken at the same time be sure photos are properly accounted for.

The primary safety measure will be erythema. It will be assessed visually without magnification using a standard dental light. Erythema (red changes) will be rated on a 1 to 3 scale, where 1 is no redness and 3 is a severe change. For subjects with more than one test tooth, scores will be averaged for all test teeth.

The Gingival Index (Löe,1967) will also be used to measure gingival inflammation.

White changes, ulceration, and staining will be secondary measures.

White changes will be rated as present or absent.

Ulceration will be rated as present or absent.

Staining (localized argyria) of the cervical gingival tissue will be rated as present or absent. The perioral area will also be assessed for argyria, present or absent.

Quality Assurance: There will be two examiners (Drs. Roccio Lazio and Shirley Rivera, who will have no role in any other aspect of the study and will be blind to study aims and group assignment. The examiners will be trained clinically to assess sensitivity and for the safety assessment, using standard photographs. As part of the training each examiner will rate 10 patients who are not part of the randomized study, and the intraclass correlation (ICC) will be calculated. Each examiner will test each patient. Each examiner will rate the gingival tissues for erythema, white changes, ulceration and staining and also take a clinical photograph of the gingival tissue at each examination.

Training for rating erythema: Trainees will view standard photographs showing no redness, some redness, and severe redness. They will each then examine and rate all 10 training patients independently, chosen to represent a range of severity. They will be allowed to refer to the standard photos during the rating. The intraclass correlation will be calculated for the two examiners. Examiners will be trained to achieve agreement with ICC=0.8 or better

Training for Gingival Index: Examiners will be instructed clinically on the GI. Then each will assess bleeding around the premolars in each of 5 patients chosen randomly from the 10 to be assessed. Scores will be calculated and the Wkappa calculated for the two examiners. Examiners will be trained to achieve agreement with ICC=0.8 or better

An independent examiner, Dr. Tar Chee Aw, who will be blind to the study conditions, will separately rate the post-treatment photographs of the gingival tissues for erythema, white changes, ulceration and staining in the same manner as the clinical examiner but without access to the earlier ratings. The photographs will be masked to avoid bias from tooth staining and will be presented to the examiner in random order. The intraclass correlation (ICC) to assess between-examiner reliability will be calculated.

Case-report forms have been developed and local staff trained in their use. Original forms and photographs will be kept in a site notebook, stored in a locked cabinet, and be readily available for audit. All entries will be in black ink, signed and dated. Copies will be made and sent to the data coordinating center at the University of Washington for entry and analysis.

Clinical Procedure: All tooth surfaces that meet the entry criteria will be treated in an individual's mouth up to a limit of 3 surfaces per patient. All the surfaces in an individual will receive the same treatment. The surface will be isolated with a cotton roll and then will be gently dried with cotton gauze. A disposable dental microbrush (Kerr Quiktips) will be dipped in a small drop of diammine silver fluoride or water and then applied to the surface for 1 second, as is done clinically. Then the surface will be gently air-dried. Then the procedure will be repeated.

At this point each of the two examiners, blind to the aims of the study and treatment condition, will begin the assessment for both sensitivity and safety. The follow-up assessment will be conducted at 24 hours and again at 1 week.

Analysis:

The data from the two sites will be analyzed separately to demonstrate the treatment effect on tooth pain. To confirm reduction in pain (sensitivity, the clinical indication), average difference scores between pretreatment and post- treatment VAS scores for each individual will be calculated for each time point (immediately after treatment, and 24 hours and 1 week after treatment) and t-tests will be used to compare changes. The primary end point will be at 1 week. GEE linear regression will be used in a secondary analysis to compare the reduction in pain across the three time points, where the outcome is sensitivity at the three time points, the baseline pain is a covariate, and robust standard errors are used to account for multiple observations per subject. In addition, separate analyses of covariance will be done at each time point to compare the reduction in pain due to the active treatment between the two study sites, where the outcome is the pain a particular time point, baseline pain is entered as a covariate, and treatment and site, as well as an treatment group by site interaction, are entered as factors.

Fisher's Exact Test will be used to assess whether there are more subjects with erythema score >1 in the diammine silver fluoride group versus the control group. (The tests will be conducted separately at each time period, immediately after treatment, at 24 hours and 1 week.) Initially tests will be conducted separately by site, then by combining both sites to increase the statistical power to detect differences in the safety measures. The primary end point will be assessed at 24 hours. A t-test test will assess any differences in Gingival Index. Any white changes, ulceration and staining (argyria) will be reported.

Power Analysis:

The data from the two sites will be analyzed separately, and power is described for the separate site analyses.

Reduction in Tooth Sensitivity (clinical indication): The primary end point will be assessed at 7 days post-treatment. In a similar desensitization study comparing several devices including the predicate device (Ritter et al., 2006, paper appended) pain on air-blast reports for Duraphat dropped from 36.9 (SD=26.2) at baseline to 20.8 (SD=4.3) at 24 weeks post-treatment. We expect a similar or much larger drop after 7 days with DASF, based on unpublished work from the University of Hong Kong (data appended) and little or no drop from the application of sterile water. The Hong Kong data suggest we will achieve a much greater reduction in tooth sensitivity than observed in the Ritter study. Thus a sample size of 31 in a group will allow detection of effect size from 0.64 (calculated from the Duraphat work) upwards with an alpha of 0.05 and power of 0.8 (one-sided test, online calculator: http://www.danielsoper.com/statcalc/calc47.aspx). To increase the statistical power to detect smaller differences, the outcome data will also be analyzed for both sites combined.

We expect no (or at least very low) attrition over the short time period of the study, but to account for possible attrition, the sample size will be inflated to 144 or 72 per site.

Based on Fisher's Exact Test and separate analyses by site with only 25 subjects per group the power is 86% to detect a difference in the proportion of subjects with a gingival inflammation score >1 of 10 out of 25 (40%) versus 1 out of 25 (4%) and 85% to detect a difference of 8 out of 25 (32%) versus 0 out of 25 (0%). To increase the statistical power to detect smaller differences, the safety outcomes will be also analyzed for both sites combined. Based on Fisher's Exact Test with 50 subjects per group the power is 84% to detect a difference of 9 out of 50 (18%) versus 1 out of 50 (2%) and 80% to detect a difference of 4 out of 50 (8%) versus 0 out of 50 (0%) (Bertil Olofosson, StudySize, Version 2.0.4, CreoStat HB, 2007). Note: no recent studies have reported any gingival inflammatory changes, nor do we expect to see any.

ELIGIBILITY:
Inclusion Criteria:

* To be included the subject must have at least one vital maxillary or mandibular cuspid or premolar with a cervical defect on the buccal surface and clinical hypersensitivity in response to air with a score not less than 15 on the VAS for pain (described below).
* The individual will have generally healthy gum tissue surrounding this tooth and no ulceration, and no leukoplakia (white changes) in this gingival tissue.

Exclusion Criteria:

* Excluded will be subjects who are using any type of commercially available tooth desensitizer, have received a fluoride varnish treatment within the last month, or who are taking prescription medications of any kind, are taking aspirin or nonsteroidal anti-inflammatory drugs habitually, and women who are pregnant.
* Individuals using smokeless tobacco will be excluded. Individuals with known sensitivity to silver or other heavy-metal ions will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Erythema | 1 week
Sensitivity | 1 week
Gingival index | 1 week

SECONDARY OUTCOMES:
white changes | 1 week
ulceration | 1 week
staining | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Principal Investigator — University of Washington; Jorge L Castillo, DDS MS, Principal Investigator — Universidad Peruana Cayetano Heredia
Locations (2):
- Peru (2):
  - Universidad Andina del CUsco, Cusco, Departamento de Cusco
  - Universidad Peruana Cayetano Heredia, Lima, Lima Province